CLINICAL TRIAL: NCT06145607
Title: A Phase 1 Study to Evaluate Safety, Tolerability, and Food-Effect Following Administration of ABBV-CLS-7262 in Healthy Volunteers
Brief Title: A Phase 1 Study Assessing the Effect of Food on the Pharmacokinetics of ABBV- CLS-7262
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calico Life Sciences LLC (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M24-851
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Food effect; Pharmacokinetics

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Period 1, 2 and 3 ABBV-CLS-7262 (Experimental): * Participants will receive ABBV-CLS-7262 administered under fasted conditions.
  * Participants will receive ABBV-CLS-7262 administered under fed conditions (high-fat/high-calorie breakfast).
  * Participants will receive ABBV-CLS-7262 administered with applesauce.
  Interventions: Drug: ABBV-CLS-7262

INTERVENTIONS:
Drug: ABBV-CLS-7262 — ABBV-CLS-7262

SUMMARY:
This study is a randomized, three period, six sequence, single dose crossover design with ABBV-CLS-7262 in healthy adult subjects.

DETAILED DESCRIPTION:
On Day 1 of each period, subjects will receive a single oral dose of ABBV-CLS-7262 administered according to the food regimen assigned. There will be a 4-day washout period between doses. Food regimens include administration after fasting, following a high-fat/high-calorie meal, or with apple sauce. Upon completion each subject will have taken a total of three doses of ABBV-CLS-7262, with one dose administered with each food regimen.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers in general good health.
* Must voluntarily sign and date an informed consent, approved by an independent ethics committee (IEC)/institutional review board (IRB), prior to the initiation of any screening or study-specific procedures.
* Individuals between 18 and 55 years of age inclusive at the time of screening.
* Body Mass Index (BMI) is ≥ 18.0 to ≤ 32.0 kg/m2.
* All male subjects who are sexually active and not surgically sterilized must agree to use an acceptable contraceptive method. Additionally, male subjects must agree to not donate sperm during the study until 30 days after the final dose of study drug.
* All female subjects who are sexually active and of childbearing potential must agree to use a highly effective contraceptive method. Additionally, female subjects must agree to not donate eggs during the study and for 30 days after the final dose of study drug.

Exclusion Criteria:

* Subject who, in the opinion of the investigator, is incapable of completing study-required visits and procedures
* Pregnant or breastfeeding.
* Treatment with any other investigational treatment within 30 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics following a single oral dose of ABBV-CLS-7262 taken with or without food. | Approximately Two Weeks
  Maximum Plasma Concentration [Cmax]; Area under the Curve (AUC)
To assess the pharmacokinetics following a single oral dose of ABBV-CLS-7262 administered with or without applesauce. | Approximately Two Weeks
  Maximum Plasma Concentration [Cmax]; Area under the Curve (AUC)

SECONDARY OUTCOMES:
Safety and Tolerability | Approximately Six Weeks
  Number of patients with treatment-related adverse events as assessed by NCI CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- AbbVie Clinical Pharmacology Research Unit (ACPRU), Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No